CLINICAL TRIAL: NCT04844632
Title: COVID19 Vaccination: Clinical, Laboratory and Cellular Monitoring
Acronym: SAPIENZAVAX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Stefania Basili, Full Professor, University of Roma La Sapienza
Other Study IDs: COVID19 vaccination_Sapienza
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Health Care Utilization; Health Care Associated Infection
Keywords: Covid19; Vaccine
MeSH Terms: conditions — Patient Acceptance of Health Care; Cross Infection; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Vaccine anti-Covid19 — Vaccination with AstraZeneca or Pfizer-Biontech anti-Covid19 vaccine

SUMMARY:
Primary objective:

1. Monitor adverse events (Adverse Event Following Immunization - AEFI) in vaccinated subjects and analyze the associations with: (a) demographic variables and anthropometric parameters (sex, age, BMI, etc.); (b) socioeconomic-cultural variables; (c) co-morbidities.

Secondary objectives:

1. Monitor the antibody response in vaccinated subjects and analyze the associations with: (a) demographic variables and anthropometric parameters (sex, age, BMI, etc.); (b) socioeconomic-cultural variables; (c) co-morbidities.
2. Assess the quantity (antibody titer) and quality of the anti-Spike immune response induced by vaccination.
3. Evaluate the dynamics of the infection and the protective efficacy of the vaccine against infection / disease by studying the incidence and titre of antibodies against Nucleoprotein (N) induced by natural infection;
4. Evaluate the neutralizing capacity of sera vs. a panel of sera selected and analyzed in house and in in vitro microneutralization systems with live virus;
5. To evaluate the cell-mediated immune response (CMI) to vaccination against SARS-CoV-2 in a subgroup of vaccinees.

Methodology:

1. Administration at baseline of a questionnaire for the collection of clinical data.
2. Perform a blood sample to measure antibody response in vaccinated subjects
3. Administer a questionnaire to evaluate adverse events after vaccination
4. Reassess the antibody response 1 month after complete vaccination and 6 and 12 months after the start of vaccination
5. An antibody assay will be drawn in a subgroup before subjecting the subject to the vaccine.
6. In a subgroup, the blood collected will also be collected in a heparinized tube for the study of cell-mediated immunity.
7. In the event that a subject participating in the study presents during the course of the observation the positivity for the molecular research of SARS-CoV-2 RNA to the oro-nasopharyngeal swab, a new sample will be performed and sent to the Istituto Superiore di Sanità for the search for viral variants.

ELIGIBILITY:
Inclusion Criteria:

All subjects vaccinated or to be vaccinated at the AOU Policlinico Umberto I and who will agree to join the study.

Exclusion Criteria:

All subjects who refuse to give consent or who have contraindications to vaccination.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subjects (age> 18) booked for anti-SARS-CoV-2 vaccination at the AOU Policlinico Umberto I.
  Subjects will include healthcare personnel, medical students and university staff recruited from Sapienza University of Rome and Umberto I university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-21 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Following Immunization - AEFI | 12 months from immunization
  Adverse events (Adverse Event Following Immunization - AEFI) monitoring in vaccinated subjects and analyze associations with: (a) demographic variables and anthropometric parameters (sex, age, BMI, etc.); (b) socioeconomic-cultural variables; (c) co-morbidities.

SECONDARY OUTCOMES:
Antibody response in vaccinated subject | 1, 3, 6, 12 months from immunization
  To monitor the antibody response in vaccinated subjects and analyze the associations with: (a) demographic variables and anthropometric parameters (sex, age, BMI, etc.); (b) socioeconomic-cultural variables; (c) co-morbidities.
Anti-Spike immune response | 1, 3, 6, 12 months from immunization
  Assess the quantity (antibody titer) and quality of the anti-Spike immune response induced by vaccination.
Anti- Nucleoprotein (N) induced by natural infection evaluation | 1, 3, 6, 12 months from immunization
  To assess the dynamics of the infection and the protective efficacy of the vaccine against infection / disease by studying the incidence and titre of antibodies against Nucleoprotein (N) induced by natural infection;
Neutralizing capacity of sera | 1, 3, 6, 12 months from immunization
  to evaluate the neutralizing capacity of sera vs. a panel of sera selected and analyzed in house and in in vitro microneutralization systems with live virus
Cell-mediated immune response | Time 0 (before immunization) 3, 10, 21, 30 days; 1, 3, 6 months from immunization
  To evaluate the cell-mediated immune response (CMI) to vaccination against SARS-CoV-2 in a subgroup of vaccinees.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Umberto I, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Capozzi A, Riitano G, Recalchi S, Manganelli V, Longo A, Falcou A, De Michele M, Garofalo T, Pulcinelli FM, Sorice M, Misasi R. Antiphospholipid antibodies in patients with stroke during COVID-19: A role in the signaling pathway leading to platelet activation. Front Immunol. 2023 Mar 2;14:1129201. doi: 10.3389/fimmu.2023.1129201. eCollection 2023. PMID 36936925